CLINICAL TRIAL: NCT02120157
Title: Pediatric Blood & Marrow Transplant Consortium (PBMTC) Phase II Myeloablative Haploidentical BMT With Post-transplantation Cyclophosphamide for Pediatric Patients With Hematologic Malignancies
Brief Title: Myeloablative Haploidentical BMT With Post-transplant Cyclophosphamide for Pediatric Patients With Hematologic Malignancies
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J13161; NA_00091665 (Other: JHM IRB)
Record Dates: First submitted 2014-04-16; First posted 2014-04-22 (Estimated); Results first posted 2019-04-18 (Actual); Last update posted 2021-11-26 (Actual); Status verified 2021-11

CONDITIONS: Myeloablative Conditioning; HLA-mismatched Bone Marrow Transplantation; Graft Survival; Transplantation, Bone Marrow
Keywords: Acute lymphoblastic leukemia; Acute myeloid leukemia; Juvenile myelomonocytic leukemia; Treatment related leukemia; Biphenotypic leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Leukemia, Myelomonocytic, Juvenile | interventions — Cyclophosphamide; Busulfan; Tacrolimus; Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Haploidentical BMT with PTCy for acute leukemias and MDS (Experimental): Patients with AML and MDS:
  Days -6 through -3: Busulfan q 5-6h IV q24h x 4 days
  Days -2 and -1: Cyclophosphamide 50mg/kg/day IV x 2 days+ Mesna 40 mg/kg/day IV
  For patients with ALL and lymphoblastic lymphoma:
  Days -5 through -4: Cyclophosphamide 50mg/kg/day IV q24h x 2 days+Mesna 40 mg/kg/day IV
  Days -3 through -1: TBI 200 Centigray (cGy) twice a day for 3 days
  All patients Day 0: Infuse unmanipulated bone marrow
  Day +3 and +4: Cyclophosphamide 50 mg/kg/day IV + Mesna 40 mg/kg IBW/day IV
  Day +5: Begin tacrolimus 0.015mg/kg IBW/dose IV over 4 hours q 12h and mycophenolate mofetil (MMF)15mg/kg po/IV tid with maximum daily dose 3 gm/day
  Day +30: Assess chimerism and disease status in bone marrow
  Day +35: Discontinue MMF
  Day +60: Assess chimerism and disease status in bone marrow
  Day 180: Discontinue tacrolimus
  Interventions: Drug: Cyclophosphamide; Radiation: TBI; Drug: Busulfan; Other: Unmanipulated Bone Marrow; Drug: Tacrolimus; Drug: Mycophenolate mofetil

INTERVENTIONS:
Drug: Cyclophosphamide — Chemotherapy administration
  Other Names: Cy
Radiation: TBI — Radiation Therapy
Drug: Busulfan — Chemotherapy Administered
  Other Names: Bu
Other: Unmanipulated Bone Marrow — Bone Marrow Transplant
Drug: Tacrolimus — Immunosuppressive Drug Administered
  Other Names: tacro
Drug: Mycophenolate mofetil — Immunosuppressive Drug Administered
  Other Names: MMF

SUMMARY:
This is a multi-institutional phase II haploidentical T cell replete bone marrow transplant (BMT) study in children with high-risk leukemia. The myeloablative conditioning regimen prescribed will be Total body irradiation (TBI)-based for lymphoid leukemia and busulfan-based for myeloid leukemia. Our goal is to establish an easily exportable, inexpensive platform for haplotransplantation that has a safety profile equivalent to matched related and unrelated BMTs. The primary objective will be to estimate the incidence of 6-month non-relapse mortality (NRM), hypothesizing that NRM is < 18%.

DETAILED DESCRIPTION:
This is a phase II prospective study designed to evaluate the incidence of 6 month non- relapse mortality, safety, and feasibility of haploidentical bone marrow transplantation (BMT) after myeloablative conditioning with post-transplant Cy. Conditioning regimens include a total body irradiation (TBI)-based prep for lymphoid leukemias and a chemotherapy based prep for myeloid leukemias.

To estimate the incidence of non-relapse mortality at 180 days following myeloablative haploidentical BMT for children and young adults with high risk hematologic malignancies.

ELIGIBILITY:
Inclusion Criteria:

* Patient age 0.5-25years
* Patients must have a first-degree related donor or half-sibling who is at minimum HLA haploidentical. The donor and recipient must be identical at at least one allele of each of the following genetic loci: HLA-A, HLA-B, HLA-Cw, HLA-DRB1, and HLA-DQB1. A minimum match of 5/10 is therefore required, and will be considered sufficient evidence that the donor and recipient share one HLA haplotype.
* An unrelated donor search is not required for a patient to be eligible for this protocol, or a donor search and donor mobilization may be abandoned if the clinical situation dictates an urgent transplant. Clinical urgency is defined as 6-8 weeks from referral to transplant or a low-likelihood of finding a matched, unrelated donor. Patients with an eligible HLA-matched RELATED should not be enrolled on this trial.
* Patients must have at least one of the following high-risk conditions listed below:
* Acute lymphocytic leukemia (ALL) in CR1* as defined by at least one of the following:

hypodiploidy, induction failure,Minimal residual disease (MRD) after consolidation

- Acute myeloid leukemia (AML) in CR1 with high risk features defined as: High allelic ratio FLT3/ITD+, Monosomy 7, Del (5q), Standard risk cytogenetics with positive minimal residual disease at the end of Induction I chemotherapy (for patients being treated on or according to Children's Oncology Group (COG) AAML1031 study who have had MRD studies sent to Seattle or performed at their local institution where the flow assay is sensitive enough to detect > 0.1% blasts)

* Acute Leukemia in 2nd or subsequent CR (CR>2)
* Mixed phenotype/Undifferentiated Leukemia in 1st or subsequent CR*
* Secondary or therapy related leukemia in CR > 1
* Natural Killer (NK) cell lymphoblastic leukemia CR > 1
* Myelodysplastic syndrome (MDS)
* Juvenile myelomonocytic leukemia (JMML) (patients are eligible if they are not eligible for COG1221 study)
* Prior transplant eligible if < 18yo, >6 months has elapsed since BMT, and patient is off immunosuppression for > 3 months with no Graft versus host disease (GVHD)
* No known active Central nervous system (CNS) involvement or extramedullary involvement by malignancy. Such disease treated into remission is permitted.
* Acute Leukemia - Remission is defined as morphology with < 5% blasts with no morphological characteristics of acute leukemia (e.g., Auer Rods) in a bone marrow with > 20% cellularity.

Exclusion Criteria:

* Poor cardiac function: left ventricular ejection fraction <45% as determined by Multigated acquisition scan (MUGA) or Echocardiogram (ECHO). For pediatric patients Left ventricular ejection fraction (LVEF) <45% or a shortening fraction below normal limits for age.
* Symptomatic pulmonary disease. Poor pulmonary function: Forced expiratory volume (FEV1), Forced vital capacity (FVC), and Diffusing capacity for carbon monoxide (DLCO) <50% predicted (corrected for hemoglobin) for patients who have not received thoracic or mantle irradiation. For patients who have received thoracic or mantle irradiation, FEV1 and FVC <70% predicted or DLCO < 50 of predicted. For children unable to perform Pulmonary function tests (PFTs) because of developmental stage pulse oximetry < 92% on Room air (RA).
* Poor liver function: bilirubin >2 mg/dl (not due to hemolysis, Gilbert's or primary malignancy). Alanine aminotransferase (ALT) or Aspartate transaminase (AST) > 3 x laboratory upper normal limits.
* Poor renal function: Creatinine >2.0mg/dl or creatinine clearance (calculated creatinine clearance is permitted) < 60 mL/min based on Traditional Cockcroft-Gault formula: 140 - age (yrs) x Smaller of Actual Weight vs. Ideal Body Weight (kg) / 72 x Serum creatinine (mg/dl) Multiply by another factor of 0.85 if female Intended for ages 18-110, serum creatinine 0.6-7 mg/dl For patients <18 years: creatinine clearance (CrCl) will be estimated by the Schwartz formula. A measured CrCl or a Glomerular filtration rate (GFR) may be substituted to determine the subject's CrCl.
* Schwartz equation: CrCl (ml/min/1.73m2)=[length (cm) x k] /serum creatinine K = 0.45 for infants 1 to 52 weeks old k = 0.55 for children 1 to 13 years old k = 0.55 for adolescent females 13-18 years old k = 0.7 for adolescent males 13-18 years old
* HIV-positive
* Positive leukocytotoxic crossmatch Specifically, complement dependent cytotoxicity and flow cytometric crossmatch assays must be negative, and the mean fluorescence intensity (MFI) of any anti-donor HLA antibody by solid phase immunoassay should be <3000. Consult with PI for the clinical significance of any anti-donor antibody.
* Women of childbearing potential who currently are pregnant (HCG+) or who are not practicing adequate contraception or who are breastfeeding
* Uncontrolled viral, bacterial, or fungal infections (currently taking medication and have progression of clinical symptoms)
* Patients with symptoms consistent with Respiratory syncytial virus (RSV), influenza A, B, or parainfluenza at the time of enrollment will be assayed for the above viruses and if positive are not eligible for the trial until they are no longer symptomatic (patients may have continued assay positivity for a period of time post resolution of symptoms secondary to the nature of the assay

Ages: 6 Months to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 35 (Actual)
Dates: Start 2015-07-02 (Actual); Primary Completion 2018-06-15 (Actual); Study Completion 2020-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Heather Symons, MD, MHS, Principal Investigator — SKCCC Johns Hopkins Hospital
Locations (9):
- United States (7):
  - Children's Hospital of Colorado, Aurora, Colorado
  - Nemours Alfred I. DuPont Hospital for Children, Wilmington, Delaware
  - All Children's Hospital Johns Hopkins Medicine, St. Petersburg, Florida
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Washington University in St. Louis, St Louis, Missouri
  - Levine Cancer Center, Charlotte, North Carolina
  - Medical University of South Carolina, Charleston, South Carolina
- Canada (2):
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - Hospital for Sick Children, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fierro-Pineda JC, Tsai HL, Blackford A, Cluster A, Caywood E, Dalal J, Davis J, Egeler M, Huo J, Hudspeth M, Keating A, Kelly SS, Krueger J, Lee D, Lehmann L, Madden L, Oshrine B, Pulsipher MA, Fry T, Symons HJ. Prospective PTCTC trial of myeloablative haplo-BMT with posttransplant cyclophosphamide for pediatric acute leukemias. Blood Adv. 2023 Sep 26;7(18):5639-5648. doi: 10.1182/bloodadvances.2023010281. PMID 37257193

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Three patients screen failed due to: One patient could not report on whether the marrow is cellular or at least 20 percent cellularity, one patient had poor liver function, and the one patient's Alanine aminotransferase (ALT) was over the study limit.
Groups:
- Haploidentical BMT With PTCy for Acute Leukemias and MDS: Patients with acute myelogenous leukemia (AML) and myelodysplastic syndrome (MDS):
  Days -6 through -3: Busulfan q 5-6h IV q24h x 4 days Days -2 and -1: Cyclophosphamide 50mg/kg/day IV x 2 days+ Mesna 40 mg/kg/day IV
  For patients with acute lymphocytic leukemia (ALL) and lymphoblastic lymphoma:
  Days -5 through -4: Cyclophosphamide 50mg/kg/day IV q24h x 2 days+Mesna 40 mg/kg/day IV Days -3 through -1: total body irradiation (TBI) 200 Centigray (cGy) twice a day for 3 days All patients Day 0: Infuse unmanipulated bone marrow Day +3 and +4: Cyclophosphamide 50 mg/kg/day IV + Mesna 40 mg/kg IBW/day IV Day +5: Begin tacrolimus 0.015mg/kg IBW/dose IV over 4 hours q 12h and mycophenolate mofetil (MMF)15mg/kg po/IV tid with maximum daily dose 3 gm/day Day +30: Assess chimerism and disease status in bone marrow Day +35: Discontinue MMF Day +60: Assess chimerism and disease status in bone marrow Day 180: Discontinue tacrolimus Cyclophosphamide: Chemotherapy administration TBI: Radiation Therapy Busulfan: Chemotherapy Administered Unmanipulated Bone Marrow: Bone Marrow Transplant Tacrolimus: Immunosuppressive Drug Administered Mycophenolate mofetil: Immunosuppressive Drug Administered
Period: Overall Study
Arm/Group | Haploidentical BMT With PTCy for Acute Leukemias and MDS
Started | 32
Completed 180 Days | 30
Completed | 24
Not Completed | 8
Not completed — Death | 8

BASELINE CHARACTERISTICS:
Arm/Group | Haploidentical BMT With PTCy for Acute Leukemias and MDS
Number analyzed (Participants) | 32
Age, Continuous [Median (Full Range); unit: years] | 12 [1 to 23]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11
  Not Hispanic or Latino | 21
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 18
  More than one race | 4
  Unknown or Not Reported | 2
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 7
  United States | 25

OUTCOME MEASURES:

1. Primary Outcome: Cumulative Incidence of Non-relapse Mortality
Description: Cumulative incidence (measured as a percentage) of non-relapse mortality at 180 days following myeloablative, Human Leukocyte Antigen (HLA)-mismatched bone marrow transplant (BMT) for patients with high risk hematologic malignancies.
Time Frame: Day 180
Measure: Number; unit: percent
Arm/Group | Haploidentical BMT With PTCy for Acute Leukemias and MDS
Number analyzed (Participants) | 32
percent | 0

2. Secondary Outcome: Number of Participants With Donor Cell Engraftment
Description: Number of Participants with Donor Cell Engraftment at Day 60 following myeloablative, HLA-mismatched BMT.
Time Frame: Day 60
Measure: Count of Participants; unit: Participants
Groups:
- Haploidentical BMT With PTCy for Acute Leukemias and MDS: Patients with AML and MDS:
  Days -6 through -3: Busulfan q 5-6h IV q24h x 4 days Days -2 and -1: Cyclophosphamide 50mg/kg/day IV x 2 days+ Mesna 40 mg/kg/day IV
  For patients with ALL and lymphoblastic lymphoma:
  Days -5 through -4: Cyclophosphamide 50mg/kg/day IV q24h x 2 days+Mesna 40 mg/kg/day IV Days -3 through -1: TBI 200 Centigray (cGy) twice a day for 3 days All patients Day 0: Infuse unmanipulated bone marrow Day +3 and +4: Cyclophosphamide 50 mg/kg/day IV + Mesna 40 mg/kg IBW/day IV Day +5: Begin tacrolimus 0.015mg/kg IBW/dose IV over 4 hours q 12h and mycophenolate mofetil (MMF)15mg/kg po/IV tid with maximum daily dose 3 gm/day Day +30: Assess chimerism and disease status in bone marrow Day +35: Discontinue MMF Day +60: Assess chimerism and disease status in bone marrow Day 180: Discontinue tacrolimus Cyclophosphamide: Chemotherapy administration TBI: Radiation Therapy Busulfan: Chemotherapy Administered Unmanipulated Bone Marrow: Bone Marrow Transplant Tacrolimus: Immunosuppressive Drug Administered Mycophenolate mofetil: Immunosuppressive Drug Administered
Arm/Group | Haploidentical BMT With PTCy for Acute Leukemias and MDS
Number analyzed (Participants) | 32
Participants | 27

3. Secondary Outcome: Cumulative Incidence of Acute Graft Versus Host Disease (GVHD) Grades 2-4 and Grades 3-4
Description: Cumulative incidence (measured as a percentage) of acute GVHD grades 2-4 (overall) and grades 3-4 (severe).
Time Frame: 100 days
Measure: Number; unit: percent
Arm/Group | Haploidentical BMT With PTCy for Acute Leukemias and MDS
Number analyzed (Participants) | 32
percent
  Grades 2-4 | 10
  Grades 3-4 | 0

4. Secondary Outcome: Cumulative Incidence of Chronic GVHD
Description: Cumulative incidence (measured as a percentage) of chronic graft versus host disease (GVHD).
Time Frame: 2 years
Measure: Number; unit: percent
Arm/Group | Haploidentical BMT With PTCy for Acute Leukemias and MDS
Number analyzed (Participants) | 32
percent | 11

5. Secondary Outcome: Primary and Secondary Graft Failure
Description: Incidence (measured as a percentage) of primary and secondary graft failure.
Time Frame: 2 years
Measure: Number; unit: percentage of graft failure
Arm/Group | Haploidentical BMT With PTCy for Acute Leukemias and MDS
Number analyzed (Participants) | 32
percentage of graft failure
  Primary | 16
  Secondary | 0

6. Secondary Outcome: Steroid and Non-steroid Immunosuppressants
Description: Number of participants who used steroid and non-steroid immunosuppressants to treat GVHD.
Time Frame: Two Years
Measure: Count of Participants; unit: Participants
Arm/Group | Haploidentical BMT With PTCy for Acute Leukemias and MDS
Number analyzed (Participants) | 32
Participants
  Steroid immunosuppressants | 4
  Non-steroid immunosuppressants | 2

7. Secondary Outcome: Steroid and Non-steroid Immunosuppressants Use Duration
Description: Duration of use of steroid and non-steroid immunosuppressants (in months) to treat GVHD.
Time Frame: Two Years
Population: Four participants used immunosuppressants. Four used steroids and 2 of the 4 also used non-steroid. Duration of use for 3 participants using steroids was not recorded. One participant using non-steroid was not recorded.
Measure: Number; unit: months
Arm/Group | Haploidentical BMT With PTCy for Acute Leukemias and MDS
Number analyzed (Participants) | 2
months
  Steroid immunosuppressants: number analyzed (Participants) | 1
  Steroid immunosuppressants | 18
  Non-steroid immunosuppressants: number analyzed (Participants) | 1
  Non-steroid immunosuppressants | 19

8. Secondary Outcome: Survival
Description: Estimate incidence of overall survival (OS), progression-free survival (PFS), disease-free survival (DFS), event-free survival, and relapse-free GVHD-free survival (GRFS) in patients receiving myeloablative, HLA-mismatched BMT for patients with high risk hematologic malignancies at 1 year. Incidence as a percentage.
Time Frame: up to 1 years
Measure: Number; unit: percent
Arm/Group | Haploidentical BMT With PTCy for Acute Leukemias and MDS
Number analyzed (Participants) | 32
percent
  overall survival (OS) | 77
  progression-free survival (PFS) | 68
  disease-free survival (DFS) | 68
  event-free survival | 68
  Relapse-free GVHD-free survival (GRFS) | 65

9. Secondary Outcome: Survival
Description: Estimate incidence of overall survival (OS), progression-free survival (PFS), disease-free survival (DFS), event-free survival, and relapse-free GVHD-free survival (GRFS) in patients receiving myeloablative, HLA-mismatched BMT for patients with high risk hematologic malignancies at 2 years. Incidence as a percentage.
Time Frame: up to 2 years
Measure: Number; unit: percent
Arm/Group | Haploidentical BMT With PTCy for Acute Leukemias and MDS
Number analyzed (Participants) | 32
percent
  overall survival (OS) | 73
  progression-free survival (PFS) | 64
  disease-free survival (DFS) | 64
  event-free survival | 64
  Relapse-free GVHD-free survival (GRFS) | 52

10. Secondary Outcome: Immune Reconstitution
Description: Characterize immune reconstitution post myeloablative haploidentical BMT with Post transplantation cyclophosphamide (PT/Cy).
Time Frame: Two Years
Population: Blood samples collected were not analyzed due to lack of funding. No data was generated.
Arm/Group | Haploidentical BMT With PTCy for Acute Leukemias and MDS
Number analyzed (Participants) | 0

11. Secondary Outcome: Time to Neutrophil and Platelet Recovery
Description: Time to neutrophil and platelet recovery in median days
Time Frame: 100 days
Measure: Median (Full Range); unit: days
Arm/Group | Haploidentical BMT With PTCy for Acute Leukemias and MDS
Number analyzed (Participants) | 32
days
  neutrophil | 22 [14 to 58]
  platelet | 21 [12 to 44]

12. Secondary Outcome: Incidence of Donor Cell Engraftment
Description: Incidence of donor cell engraftment measured as the percentage of donor cell engraftment.
Time Frame: 60 days
Measure: Number; unit: percentage of donor cell engraftment
Arm/Group | Haploidentical BMT With PTCy for Acute Leukemias and MDS
Number analyzed (Participants) | 32
percentage of donor cell engraftment | 84

ADVERSE EVENTS:
Time Frame: Adverse event data was collected up to 180 days after transplantation. Mortality was observed for up to 2 year post-intervention.
Description: Adverse events reported at each visit during time at transplant center and up to 180 days post-transplantation.
Arm/Group | Haploidentical BMT With PTCy for Acute Leukemias and MDS
All-Cause Mortality (participants affected / at risk) | 8/32
Serious Adverse Events (participants affected / at risk) | 14/32
Other Adverse Events (participants affected / at risk) | 13/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Haploidentical BMT With PTCy for Acute Leukemias and MDS (N=32)
Fever (General disorders) | 3 (3)
Veno-occlusive Disease/ Hepatic Sinusoidal Obstruction Syndrome (Hepatobiliary disorders) | 4 (4)
Graft Failure (Surgical and medical procedures) | 3 (3)
Acute GVHD (Surgical and medical procedures) | 1 (1)
Broviac Cather Infection (Infections and infestations) | 1 (1)
Intracranial Hemorrhage (Blood and lymphatic system disorders) | 1 (1)
Cystitis (Renal and urinary disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Haploidentical BMT With PTCy for Acute Leukemias and MDS (N=32)
Anemia (Blood and lymphatic system disorders) | 4 (20)
Anorexia (Metabolism and nutrition disorders) | 4 (4)
Diarrhea (Gastrointestinal disorders) | 8 (10)
Fever (General disorders) | 5 (6)
Hypertension (Vascular disorders) | 3 (4)
Hypokalemia (Metabolism and nutrition disorders) | 4 (4)
Hypomagnesemia (Metabolism and nutrition disorders) | 5 (5)
Oral Mucositis (Gastrointestinal disorders) | 11 (13)
Nausea (Gastrointestinal disorders) | 4 (5)
Neutrophil Count Decreased (Investigations) | 2 (8)
Platelet Count Decreased (Investigations) | 3 (27)
Vomiting (Gastrointestinal disorders) | 8 (11)
White Blood cells decreased (Investigations) | 3 (19)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-04-20): https://cdn.clinicaltrials.gov/large-docs/57/NCT02120157/Prot_SAP_001.pdf